CLINICAL TRIAL: NCT04570215
Title: Digital Interventions in Neuro-Rehabilitation: A Small Scale Randomised Clinical Trial to Test a Web-based Therapy Application for People With Naming Difficulties With Mild- Moderate Dementia (Gotcha!).
Brief Title: Digital Interventions in Neuro-Rehabilitation: Gotcha!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18/0071
Record Dates: First submitted 2020-05-29; First posted 2020-09-30 (Actual); Results first posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Dementia; Alzheimer Disease; Anomia
Keywords: Digital Therapy; Digital intervention; Therapy app
MeSH Terms: conditions — Dementia; Alzheimer Disease; Anomia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gotcha! Therapy Application (Active Comparator): Participants will receive the Gotcha therapy daily for six weeks.Participants are required to use the app everyday for a maximum of 45 minutes. After this time they enter a twelve week block with no therapy or maintenance of therapy (see Gotcha maintenance arm).
  This aim of this arm is to invesitgate the efficacy of the Gotcha therapy for proper-noun anomia in mild-moderate patients with dementia (Alzheimer's disease, vascular dementia and mixed)
  Interventions: Other: Gotcha! Therapy application
- Gotcha! Therapy Application: Maintenance (Active Comparator): Participants will receive the Gotcha therapy for six weeks as described in the Gotcha arm. After this time they enter a twelve week block of maintenance of therapy gains made in the initial six week therapy block.
  The maintenance block consists of a weekly test of the Gotcha outcome measure to monitor the therapy gains made during the therapy block. If any previously correctly named person is incorrectly named during these weekly tests then the participant must complete a 'top-up' therapy session. They will then be tested again the following week.
  The aim of this arm is to compare Gotcha maintenance with Gotcha, to see if extra testing and therapy is required to maintain gains made during an initial intense therapy block.
  Interventions: Other: Gotcha! Therapy application; Other: Gotcha Therapy application: Maintenance

INTERVENTIONS:
Other: Gotcha! Therapy application — Gotcha! will provide an app-based therapy for people with dementia who have difficulty naming people they know well.
  The therapy element works via mass practice and feedback to the users on a trial-by-trial basis. The DNI is very simple in a way; it just presents a long series of pictures for users to name. This DNI will use speech recognition (SR) software in order to make a binary decision as to whether the user said the correct word or not. This affects what the next trial (object to name) is and what auditory cue (if any) is provided the next time the user has to name the same item.
  Other Names: Gotcha!
Other: Gotcha Therapy application: Maintenance — Gotcha! Maintenance therapy is identical to Gotcha! but takes place over a longer period of time in an attenuated form.
  Other Names: Gotcha Maintenance
  Arms: Gotcha! Therapy Application: Maintenance

SUMMARY:
Aims and background Everyone forgets the names of people they should know at times. Having dementia makes this problem worse. People with dementia have told expressed they forget the names of people they care about and this can be upsetting and embarrassing.

However, evidence shows that if people get enough practice, they can re-learn these names. The investigators, along with people with dementia and their carers, have created a fun therapy for people to get lots of practice so they can remember the names of people that are important to them.

The main aim of the study is:

To prove that Gotcha! therapy can help people with dementia to improve their ability to remember names.

Another aim is:

To find out if using the therapy is related to any changes in the brains of people with dementia.

Design and methods Participants are provided with a computer tablet to practise at home. Participants are required to think of 6-10 familiar people (family and friends) whose names they forget and want to remember better.

Participants also need to practise every day for about 30 minutes over a 6 week period so they get a large amount of therapy.

Participants will have 7 testing appointments over 12 months. At three of these appointments participants will need to have a brain scan. These scans are carried out by trained University College London professionals and will take no longer than 30 minutes each.

For the appointments where participants do not need to have a brain scan home testing can be arranged.

The investigators organise and pay for all journeys to and from University College London.

Participants

Participants can get involved in our research if they:

* Have ever experiences seeing a familiar person but can't remember their name
* Have a diagnosis of dementia (Alzheimer's disease or mixed dementia).
* Want to be part of an important and exciting research journey. Unfortunately a diagnosis of other any other types of dementia not mentioned above is not suitable for this study

Patient and Public involvement The investigators have engaged with people from the Alzheimer's Society and local dementia carers groups, run many focus groups and interviewed people with dementia and their carers to co-design the therapy.

At the end of our research participants are invited to University College London to learn about the results of the study.

DETAILED DESCRIPTION:
Background

The number of people with dementia in the UK is forecast to increase by 40% over the next 12 years and 156% over the next 38 years (Prince et al., 2014). People with all stages of Alzheimer's disease (AD) report forgetting even very familiar people's names, which patients find annoying and embarrassing (Werner, 2004). This therapy speaks to the James Lind Alliance's dementia top priority, "What are the most effective components of care that keep a person with dementia as independent as they can be at all stages of the disease in all care settings?" Several case studies and one group study have shown that patients with AD can significantly improve proper name recall with training; the effects last months after training is completed (Clare et al., 2002). Given the prevalence of mobile phone technology with inbuilt cameras and the rapid rise in usage in the 64-74 year old bracket, the investigators will develop a name-training intervention that allows people with proper name recall impairments to take pictures of and add the name of people that they wish to name. The app will include voice recognition software so that our bespoke adaptive algorithm (developed with Prof Mark Huckvale at UCL) will be able to adaptively cue users depending on their speech output.

Gotcha! will provide an app-based therapy for people with dementia who have difficulty naming people they know well.

This Digital Neuro Intervention (DNI) will provide the opportunity for the necessary increased rehabilitation to help people recover lost naming function. This will alleviate NHS Speech and Language Therapist (SALT) time and put users in control of when and where they carry out practice-based language therapy.

Identification and description of the Investigational Device

Purpose Gotcha! will provide an app-based therapy for people with dementia who have difficulty naming people they know well.

What does it do? The therapy element works via mass practice and feedback to the users on a trial-by-trial basis. The DNI is very simple in a way; it just presents a long series of pictures for users to name. This DNI will use speech recognition (SR) software in order to make a binary decision as to whether the user said the correct word or not. This affects what the next trial (object to name) is and what auditory cue (if any) is provided the next time the user has to name the same item.

*The speech will be recorded on the device but no other identifiable information will be stored on it. When the participant finishes the trial, the investigators will delete all information on the device.

What is the clinical trial design? A small, well-defined sample of patients with the potential to benefit from the DNI will be recruited. The main outcome measure is whether the DNI is effective at improving naming impairments. This comparison is within-subject and is achieved by comparing post-therapy measures to multiple baseline measures. The investigators are also comparing two different versions of the therapy (a between group comparison) to answer our secondary question of whether the therapy can be optimised. Outcome measures will be collected by the research team using a variety of standardized and non-standardized tests of language and cognition.

The DNI will be introduced to the participant when attending a testing session. One of the research team will explain how to use the DNI, provide instructions for the user, and give some time for practice items. When confident that the participant can use the DNI independently, the participant will take the device home and continue their therapy (suggested therapy time is 5-10 hours per week) which will be simultaneously monitored by the research team. The research team will also check in on the participant weekly to trouble shoot any difficulties they may have (whether motivational or technical). When the participant has completed the therapy block, the investigators will invite them in again for testing and they will return the mobile device with the DNI on it. The participants who continue to receive standard care during the therapy block will be asked to record and submit details to the research team.

Justification for the design of the clinical investigation Why is the research considered worth doing? Standard (face to face) Speech and Language Therapy (SALT) has a huge evidence-base but patients in the NHS have unmet therapy needs due to a lack of resources. The evidence from speech-therapy highlights the amount of time-on-task required to improve patients' ability to communicate. Naming problems are common and impact on the patients' wellbeing and social inclusion. There is also good evidence that current existing therapeutic approaches work.

In the NHS a patient with Alzheimer's Dementia are likely to receive little or no SALT. Our solution to the lack of available SALT therapy is to produce digital neuro-interventions that give patients the opportunity to practice scientifically validated, impairment based therapy when and where it suits them which gives them access to optimum therapy dose.

Therapy can be effortful for patients who can sometimes be too fatigued when the therapist comes to do their session. This digital neuro-intervention will provide optimum availability of therapy and therefore place the patient in control of how much they do. However, the therapy will be engaging through adaptive and exciting software. The adaptiveness will serve to reward the patients for their efforts without ever making them feel like they are failing. This will hopefully boost how long they spend in therapy and therefore make greater gains.

There are therapy apps available for patients but the scientific basis for them is lacking and none are targeted for proper name anomia. By using speech recognition software our intervention will be uniquely designed to be used by patients with word retrieval impairments.

What new information will the research provide? The concept of the therapy component is based on standard SALT practice and thus has a strong proof of concept basis, as do our proposed outcome measures. The novel component is packaging it in a user- friendly web-app that is designed for and by people with word-retrieval problems. The investigators will test the efficacy in a randomized-controlled trial (Phase 2). These digital neuro-interventions will be in contrast to the plethora of apps available online claiming cognitive training without having scientific proof.

The Gotcha! research study is a small-scale, randomised clinical trial for participants with mild to moderate dementia who have difficulty naming the people they know well (proper name anomia). The main research question is whether Gotcha! therapy improves participants' ability to freely name the people they know well. will test this hypothesis by assessing participants' naming abilities on two matched lists of people, half are trained and half remain untrained.

A secondary question relates to maintenance of therapy gains, to test this hypothesis two different versions of Gotcha! are compared, 'standard Gotcha!' and 'Gotcha! Maintenance'. These two versions are identical for the first block of therapy but differ thereafter in that the maintenance version continues to top up participants with brief training sessions over the next block while those in the standard group do not have any further interactions with the therapy. Participants will be randomised (using minimisation) to one of the two versions of the therapy. The main outcome measure will be a clinically relevant improvement on the naming ability of the trained items (compared to untrained control items). Secondary outcomes will include improvements in social activity and participation and participant and/or carer reported outcome measures (PROMS).

The investigators also plan to capture brain-based data (functional and structural MRI and MEG) in order to test a series of secondary hypotheses relating to both how and why the therapy may work in some participants but not others. All brain imaging will be outside of standard care for the participants and take place at UCL by trained staff.

Hypotheses and Objectives

H1-Primary:

Does Gotcha! improve naming performance on trained items?

This is a within-subject comparison. The criteria for success is a 10% (raw, or unstandardized) relative improvement in performance. This effect size was used in the recent Big Cactus study.

H2-Secondary:

Does Gotcha! maintenance keep participants at their maximum achieved level compared to standard Gotcha?

This is two factor analysis with both a within-subject factor (trained vs. untrained items) and a between-group factor (Gotcha! maintenance vs. standard Gotcha). The criteria for success is a 10% (raw, or unstandardized) relative difference in performance. This effect size was used in the recent Big Cactus study.

Primary Objective Does Gotcha! improve naming performance on trained items?

Secondary Objective(s)

The investigators aim to show that using this DNI will improve word retrieval on trained items by providing a known therapy used by SLT's through a digital app and by enabling an increased dose of therapy. However, the investigators also believe that by using this DNI and practicing every day, there will be changes in participants' brain structure and in the health of the participants and their carers.

* Does Gotcha! maintenance keep participants at their maximum achieved level compared to standard Gotcha?
* Are the therapy effects item-specific or do is there generalization to untrained items?
* Are the effects of the DNI therapy limited to the language domain alone or do they improve in other cognitive domains (e.g. sustained attention)?
* Does the DNI improve participant's social activity and participation?
* Is the DNI acceptable to participants (can they use it easily)?
* Is the DNI acceptable to participants' carers?
* Does the DNI improve carer health/well-being?
* Does the DNI have any economic benefits?
* Can baseline structural brain imaging explain participants' responses to the DNI?
* Can baseline structural brain imaging be used to predict incoming participants' response to the DNI?
* Can repeated-measures structural or functional brain imaging identify participant's brain areas that change in response to the DNI?

ELIGIBILITY:
Inclusion Criteria:

* Person with mild/moderate dementia
* Self-reported proper naming difficulty which we will then assess at Time Point 1 English as their dominant language
* Able to tolerate MRI brain scan
* Able to give informed consent
* Able to use the DNI (app)

Exclusion Criteria:

* No diagnosis of developmental language disorders
* No diagnosis of severe dementia or primary progressive aphasia
* No major co-existing neurological or psychiatric diagnosis
* No contraindications to brain scanner (e.g. the presence of ferromagnetic implants or other metallic or electronic objects in the body, weight over 24 stone, claustrophobia or pregnancy).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2024-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander P Leff, Professor, Principal Investigator — University College, London
Locations (1):
- University College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was from nine NHS Patient Identification Centres across the UK (100 screened) and two main databases: Joint Dementia Research (JDR) database and Dementias Platform UK, Great Minds (DPUK) database (462 screened). Of the 562 assessed for eligibility, 514 were excluded. Of the remaining 98, 40 declined participation and 14 were excluded for other reasons leaving 48.
Pre-assignment Details: 48 participants were recruited and entered the study, 10 dropped out (mostly due to COVID-19,), leaving 38 who completed the study. The background and results data pertain to these 38 participants.
Groups:
- Gotcha! Therapy Application: Participants will receive the Gotcha therapy for six weeks as described in the Gotcha arm. After this time they enter a twelve week block of maintenance of therapy gains made in the initial six week therapy block.
  The maintenance block consists of a weekly test of the Gotcha outcome measure to monitor the therapy gains made during the therapy block. If any previously correctly named person is incorrectly named during these weekly tests then the participant must complete a 'top-up' therapy session. They will then be tested again the following week.
  The aim of this arm is to compare Gotcha maintenance with Gotcha, to see if extra testing and therapy is required to maintain gains made during an initial intense therapy block.
Period: Overall Study
Arm/Group | Gotcha! Therapy Application
Started | 38
Completed | 38
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gotcha! Therapy Application
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.7 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Gotch! Outcome Measure [Mean (Standard Deviation); unit: percent correct] — The GOM is a free naming test using images of the participants' 6-10 personalized faces that they wanted to practice on. The test was completed in person at the main time points (T1-T5) and remotely during the weekly pre-therapy and therapy blocks. It was delivered via the app. As the number of items in the GOM varied across participants, these raw scores were converted into percentages ((correct responses/total number of stimuli)*100). The Famous Faces were tested using the same parameters at T1-T5 using a PowerPoint presentation.
  percent correct
    Familiar Faces (trained items) | 20 (6)
    Famous Faces (untrained items) | 19 (6)

OUTCOME MEASURES:

1. Primary Outcome: Gotcha! Outcome Measure
Description: The GOM is a free naming test using images of the participants' 6-10 personalized faces that they wanted to practice on. The test was completed in person at the main time points (T1-T4) and remotely during the weekly pre-therapy and therapy blocks. It was delivered via the app and consisted of the horizontally flipped versions of the photos that appeared as training items in order to reduce the effects of identity priming (Schacter, et al. 2004). The images were displayed for 6 seconds with a 2 second fade out. Responses were audio recorded and checked for accuracy with each attempt scoring either 1 or 0. As the number of items in the GOM varied across participants, these raw scores were converted into percentages ((correct responses/total number of stimuli)*100). The Famous Faces were tested using the same parameters at T1-T4 using a PowerPoint presentation.
Time Frame: T1 (baseline = initial assessment) to T4 (immediately following 6 weeks of Gotcha! therapy)
Population: The analysis is a 2*2 ANOVA. TIME (which has two levels: T1 = baseline vs. T4 = immediately post-therapy), and ITEM (Familiar Faces = Trained vs. Famous Faces = Untrained). This controls for time effects and test-retest effects. The main hypothesis is that the interaction will be significant, driven by improved naming of Trained items at T4.
Measure: Mean (95% Confidence Interval); unit: percentage
Groups:
- Familar Faces (Trained Items): Each partcipant picked between 6-10 familiar people that they wanted to improve their free naming of. They provided the photos of these people and they were uploaded to the Gotcha! app by the research team.
- Famous Faces (Unrained Items): At baseline (T1) partcipants were tested with 50 famous faces. A subgroup of these were marches 1 to 1 with the trained items. Matched on accuracy and then similar characteristics (gender, age).
Arm/Group | Familar Faces (Trained Items) | Famous Faces (Unrained Items)
Number analyzed (Participants) | 38 | 38
percentage
  T1 (Baseline) | 20 [14 to 26] | 18 [13 to 23]
  T4 (post-Gotcha! therapy) | 59 [49 to 69] | 17 [13 to 23]

ADVERSE EVENTS:
Time Frame: From T1-T5 ~36 weeks.
Arm/Group | Gotcha! Therapy Application
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38
Other Adverse Events (participants affected / at risk) | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-15): https://cdn.clinicaltrials.gov/large-docs/15/NCT04570215/Prot_SAP_000.pdf